CLINICAL TRIAL: NCT02273037
Title: The Fetal Heart Monitor Project - Human Energy to Save Lives: Intermittent Auscultation Using Handheld Doppler: a Randomized Controlled Trial Comparing Perinatal Outcomes in Uganda
Brief Title: Intermittent Auscultation Using Handheld Doppler: a Randomized Controlled Trial Comparing Perinatal Outcomes in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Diego Bassani, Epidemiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000031587
Record Dates: First submitted 2014-04-14; First posted 2014-10-23 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Stillbirth; Neonatal Death
Keywords: Labour; Birth asphyxia; Fetal Heart Rate Monitor; Doppler Fetal Heart Rate Monitor; Pinard Horn; Pediatrics; Uganda
MeSH Terms: conditions — Stillbirth; Perinatal Death; Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pinard horn (Placebo Comparator): Pinard horn (current practice) used to monitor the fetal heart rate in labour in this arm of the study.
  Interventions: Procedure: Partograph
- Fetal heart rate Doppler (Experimental): Doppler used to monitor the fetal heart rate in labour in this arm of the study.
  Interventions: Device: Fetal heart rate Doppler; Procedure: Partograph

INTERVENTIONS:
Device: Fetal heart rate Doppler — A wind-up, handheld fetal heart rate monitor Doppler developed by Power-free Education Technology Doppler (www.pet.org.za)
  Other Names: wind-up, handheld Doppler; fetal heart rate monitor; Power-free Education Technology Doppler (www.pet.org.za)
  Arms: Fetal heart rate Doppler
Procedure: Partograph — Graphical documentation of labour progress, and maternal and fetal well-being.
  Other Names: Partogram

SUMMARY:
A novel handheld Doppler has been developed which is rugged and is powered only by a hand crank. This study aims to test the use of this Doppler versus the Pinard horn to monitor the fetal heart rate in labour in a hospital setting in Uganda. The investigators propose that with its ease of use, both for the woman and midwife, midwives using the Doppler will identify more babies in need of prompt delivery and the risk of stillbirth and neonatal mortality will decline. In the research study, the investigators will compare the risk of stillbirths and neonatal mortality in two randomized groups of labouring women.

The second part of the study consists of an audit of the documentation in labour by midwives. The partograph is an uncomplicated, low cost form on which observations during labour are documented. It includes three sections of information: fetal condition, maternal condition and labour progress. Although the use of a partograph during labour is strongly recommended by the WHO, there are limited published systematic evaluations of the correct use of the tool. The investigators aim to use this randomized trial design to assess rates of intrapartum stillbirth and neonatal mortality in the first 24 hours after delivery, and assess the quality of partographs comparing two groups.

This trial will provide insights on the potential benefits of using handheld Doppler devices for intrapartum monitoring, and the audit of partograph quality will provide insights to improve care during labour. This study hypothesizes that the quality of partograph completion and of fetal heart rate monitoring may systematically differ between the Doppler and Pinard groups.

DETAILED DESCRIPTION:
1. Objectives:

   1. To evaluate the intervention of a wind-up, handheld Doppler fetal heart rate monitor (Doppler) and to identify implementation challenges;
   2. To identify process issues and the impact of the Doppler on rates of intrapartum stillbirth and neonatal deaths within 24 hours, in comparison to use of the Pinard horn (current practice);
   3. To assess the quality of partographs using a standardized scoring system to audit overall completion and quality, and fetal heart rate monitoring specifically; we will compare the audit results between partographs where monitoring was done with the Pinard horn versus the Doppler. The hypothesis being that the quality of partograph completion and of fetal heart rate monitoring may systematically differ between these two groups;
   4. To build the research capacity of Ugandan midwives by facilitating their participation in this research study.
2. Study design

   Equal randomization clinical trial to compare Pinard horn (current practice) versus Doppler (intervention) to monitor the fetal heart in labour.
3. Characteristics of the study population

   1. Number of participants Based on the results of a randomized controlled trial in urban Zimbabwe in 1994 [Mahomed, BMJ], the investigators hypothesize that use of a handheld Doppler fetal heart monitor will reduce the rate of intrapartum stillbirth by at least 30% compared to monitoring fetal heart rate with a Pinard horn. With 80% power to detect at least a 30% reduction in stillbirths with 95% confidence, 840 labouring women would need to be enrolled in each of the two comparison groups. Adding 20% to allow for losses to follow-up and statistical adjustments/stratification, 1008 labouring women are required for each comparison group.
   2. Location of the research The study will be conducted in the San Raphael of St Francis Hospital Nsambya Hospital, in Uganda. This is a general hospital and maternity located in the peri-urban region of Kampala City. It is a private not-for-profit institution with 7,500 annual deliveries. In addition, it offers training for residents, intern doctors, nurses, midwives and technicians.
4. Data analysis The investigators will review the partograph and record their findings on a tool developed for this purpose. The data that will be recorded will be of statistical nature but at the bottom of each Partograph Assessment Tool is space for qualitative comments from the reviewer. Besides date of birth and the patient file identity number no data will be recorded which can reveal the identity of the patient. This is to ensure patient privacy and confidentiality of the data, without losing the possibility to retrieve the file from medical records if needed. After recording the data on a hard copy in the hospital, the data will be entered twice into the statistical package before analysis. The information that this will give will be descriptively analysed. The proportion and incidence risk rate of participants who experience each fetal outcome under study and the mean partograph scores will be compared between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* All mothers presenting to the labour wards in labour with a singleton pregnancy above 37 completed weeks of gestation, and cephalic presentation
* All mothers admitted to the labour ward for monitoring of active phase of labour with a live intrauterine fetus

Exclusion Criteria:

* Mothers admitted to the labour wards with a pregnancy gestation age below 37 weeks
* Mothers admitted with a diagnosis of intra uterine fetal death
* Mothers presenting in second stage of labour
* Mothers with a high risk pregnancy eg pre eclampsia, ante partum hemorrhage
* Mothers being admitted for an elective caesarean section

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1987 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Bassani, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Nsambya Hospital, Kampala, Uganda

RESULTS

PARTICIPANT FLOW:
Groups:
- Pinard: Pinard Auscultation (standard of care)
- Doppler: Doppler Auscultation (Intervention)
Period: Overall Study
Arm/Group | Pinard | Doppler
Started | 987 | 1000
Completed | 979 | 992
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Delivered before monitoring initiated | 1 | 3
Not completed — Breech delivery | 2 | 3
Not completed — Multiple delivery | 2 | 2
Not completed — Other complication | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pinard: Pinard
- Doppler: Doppler
- Total: Total of all reporting groups
Arm/Group | Pinard | Doppler | Total
Number analyzed (Participants) | 979 | 992 | 1971
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 30] | 27 [24 to 30] | 27 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 979 | 992 | 1971
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 979 | 992 | 1971

OUTCOME MEASURES:

1. Primary Outcome: Stillbirth and Neonatal Death
Description: Compare the incidence of fresh stillbirth and neonatal death (within 24h of age) in the Pinard group (current practice) and the Doppler group (study intervention).
Time Frame: 0-24hour of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Pinard Horn | Fetal Heart Rate Doppler
Number analyzed (Participants) | 979 | 992
Participants | 6 | 11

2. Primary Outcome: Quality of Partograms
Description: To assess the quality of partographs using a standardized scoring system to audit overall completion and quality, and fetal heart rate monitoring specifically. The investigators will compare the audit results between partographs in the Pinard and Doppler group.
Time Frame: in labour
Reporting Status: Not Posted

3. Secondary Outcome: Identification of Abnormal Fetal Heart Rate
Description: Compare the incidence of identification of abnormal fetal heart rate in labour in the Pinard and Doppler group.
Time Frame: In labour
Measure: Count of Participants; unit: Participants
Arm/Group | Pinard | Doppler
Number analyzed (Participants) | 979 | 992
Participants | 46 | 75

4. Secondary Outcome: Cesarean Delivery (Includes Cesarean Delivery/Intra-uterine Resuscitation/Assisted Delivery)
Description: Compare the proportion of cesarean delivery between the Pinard and Doppler group.
  (Includes Cesarean Delivery/Intra-uterine Resuscitation/Assisted delivery)
Time Frame: Birth
Measure: Count of Participants; unit: Participants
Arm/Group | Pinard | Doppler
Number analyzed (Participants) | 979 | 992
Participants
  Cesarean Delivery following abnormality detection | 61 | 89
  Cesarean Delivery | 166 | 175

ADVERSE EVENTS:
Arm/Group | Pinard | Doppler
All-Cause Mortality (participants affected / at risk) | 6/979 | 11/992
Serious Adverse Events (participants affected / at risk) | 0/987 | 0/1000
Other Adverse Events (participants affected / at risk) | 0/979 | 0/992

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No